CLINICAL TRIAL: NCT00696592
Title: A Randomized, Controlled, Open Label, Phase II Study of Visudyne® Photodynamic Therapy (PDT) Combined With Bevacizumab (Avastin) vs Avastin Alone in Patients With Neovascular Age-related Macular Degeneration (AMD)
Brief Title: Photodynamic Therapy Combined With Bevacizumab vs Bevacizumab Alone for Neovascular Age-related Macular Degeneration
Acronym: ARMAST
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: new data from clinical trials
Sponsor: University of Padova (Other)
Collaborators: Department of Ophthalmology, Conegliano Hospital, Treviso, Italy (Unknown)
Responsible Party: Principal Investigator, Stefano Piermarocchi, MD, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-01-ARMAST-2007
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Age-Related Macular Degeneration; Choroidal Neovascularization; Bevacizumab; Photodynamic Therapy
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Bevacizumab; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BVZ and PDT (Experimental)
  Interventions: Drug: Bevacizumab (Avastin), Verteporfin (Visudyne)
- BVZ only (Active Comparator)
  Interventions: Drug: Bevacizumab (Avastin), Verteporfin (Visudyne)

INTERVENTIONS:
Drug: Bevacizumab (Avastin), Verteporfin (Visudyne)

SUMMARY:
This phase II study was designed to evaluate the safety, tolerability, and efficacy of bevacizumab treatment in conjunction with PDT at the low fluence rate compared with bevacizumab alone or combined with PDT at the standard fluence rate, in patients with all types of choroidal neovascularization secondary to AMD.

Hypothesis: bevacizumab in combination with PDT (low and standard fluence rate) will i) delay time to retreatment, ii) reduce the average number of treatments required compared to bevacizumab alone and iii) at low PDT fluence rate will improve long-term safety profile.

ELIGIBILITY:
Inclusion Criteria:

* All lesion subtype of CNV secondary to age-related macular.
* sub-foveal CNV.
* patients who fail to respond to Photodynamic therapy.
* patients who are not eligible for PDT (Greatest linear dimension of the lesion >/= 5400 um, CNV with hemorrhage >/= 50 % of the entire lesion, minimally classic or occult CNV with greatest linear dimension of the lesion >/= 4600 um.).
* Patients affected by Pigment Epithelium Detachment with CNV.
* Patients affected by Retinal Angiomatous Proliferation.
* Willingness and ability to participate and provide written informed consent.

Exclusion Criteria:

* Individuals with choroidal neovascularization from causes other than AMD (Myopia, Angioid Streaks).
* Any intraocular surgery within 2 months in the study eye.
* Prior retinal or vitreous surgery including posterior segment vitrectomy or scleral buckling in the study eye.
* Any significant ocular disease that has compromised or could compromise vision in the study eye.
* Prior stroke, myocardial infarction, or end-stage malignancy.
* Active hepatitis or clinically significant liver disease, renal failure.
* Any patient with recent history of new onset cardiac disease or thromboembolic CNS event in the past.
* Patients who are in an experimental therapy study or who have received experimental therapy within the last 12 weeks.
* Patients who are a poor medical risk because of other systemic diseases or active uncontrolled infections.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01-31 (Estimated); Primary Completion 2008-01-31 (Actual); Study Completion 2008-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Bevacizumab injections | One year
The mean change in best-corrected ETDRS visual acuity in the study eye | Months 6 and 12

SECONDARY OUTCOMES:
Mean change in total CNV area (Disc Areas) | Months 6 and 12
Changes of central retinal thickness measured by Optical Coherence Tomography (OCT). | Months 6 and 12
NEI VFQ-25 (vision-related quality of life) score | One year
Pelli-Robson Contrast Sensitivity Score | One year

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Piermarocchi, M.D., Principal Investigator — University of Padova
Locations (1):
- Department of Ophthalmology, University of Padova, Padua, PD, Italy